CLINICAL TRIAL: NCT01682057
Title: A Prospective, Non-Randomized, Open Label, Multi-Center Study to Evaluate the ROX Anastomotic Coupler System (ACS) in Patients With Severe Hypertension
Brief Title: A Multicenter Study to Evaluate the ROX Anastomotic Coupler System (ACS) In Patients With Severe Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ROX Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RH-01
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Hypertension
Keywords: High Blood Pressure; Hypertension; Resistant Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group A (Experimental): ROX Anastomic Coupler System (ACS) + continuing standard antihypertensive medications
  Interventions: Device: ROX ANASTOMOTIC COUPLER SYSTEM (ACS)

INTERVENTIONS:
Device: ROX ANASTOMOTIC COUPLER SYSTEM (ACS) — The ROX Anastomic Coupler (ACS) will be used to create an arteriovenous fistula in the iliac region (between the iliac artery and vein).
Device: ROX Anastomotic Coupler System (ACS)

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the ROX Anastomotic Coupler System (ACS) in patients with severe hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe hypertension must be made on the basis of current findings, medical history, and physical examination

Exclusion Criteria:

* Any serious medical condition that may adversely affect the patient's safety, limit the subject's ability to participate in the study, comply with follow-up requirements or impact the scientific integrity of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in mean office SBP | Baseline, 6 months
  Change in mean office SBP at six months as compared to Baseline

SECONDARY OUTCOMES:
Change in mean office DBP | Change in mean office DBP six months as compared to Baseline
  Change in mean office DBP at six months as compared to Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium